CLINICAL TRIAL: NCT02343926
Title: A Multicentre, National, Randomized, Parallel-group, Phase 3 Study to Compare the Efficacy and Safety of Gemigliptin and Vildagliptin as Add-on Therapy to Metformin in People With Type 2 Diabetes Inadequately Controlled With Metformin
Brief Title: Phase 3 Study to Compare the Efficacy and Safety of Gemigliptin and Vildagliptin as Add-on Therapy to Metformin in People With Type 2 Diabetes Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMIGL07185; U1111-1165-9138 (Other: UTN)
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemigliptin (Experimental): GEMIGLIPTIN LS15-0444 administered once a day for 24 weeks as add-on therapy to metformin
  Interventions: Drug: GEMIGLIPTIN LS15-0444; Drug: metformin
- Vildagliptin (Active Comparator): Vildagliptin administered twice a day for 24 weeks as add-on therapy to metformin
  Interventions: Drug: vildagliptin; Drug: metformin

INTERVENTIONS:
Drug: GEMIGLIPTIN LS15-0444 — Pharmaceutical form:tablet
  Route of administration: oral
  Other Names: Zemiglo
  Arms: Gemigliptin
Drug: vildagliptin — Pharmaceutical form:tablet
  Route of administration: oral
  Other Names: Galvus
  Arms: Vildagliptin
Drug: metformin — Pharmaceutical form:tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To compare the clinical efficacy of gemigliptin and vildagliptin as add-on therapy to metformin in terms of change in Hemoglobin A1c (HbA1c) reduction.

Secondary Objectives:

To compare the safety and tolerability of gemigliptin and vildagliptin:

* Number of patients who experience at least one episode of hypoglycemia.
* Number of patients experiencing adverse event (AE), serious adverse event (SAE).
* Assessment of patients compliance defined as number tablets returned by patients.

DETAILED DESCRIPTION:
The study consists of 2 weeks screening and 24 weeks of treatment (a total of 26 weeks).

The protocol includes a screening period of two weeks, after which they will be randomized to receive gemigliptin or vildagliptin.

Patients will be evaluated through 4 mandatory visits during the study. Visit 1: Week -2 (screening) Visit 2: Week 0 (randomization) Visit 3: Week 12 (efficacy and safety evaluation) Visit 4: Week 24 (efficacy and safety evaluation)

ELIGIBILITY:
Inclusion criteria:

* Patients with Type 2 diabetes mellitus.
* Patients inadequately controlled with metformin at the maximal effective and tolerated dose of metformin for at least 12 weeks or who are on a stable dose of ≥1500 mg daily for a minimum of ≥4 weeks prior to study entry.
* Signed informed consent obtained prior to any study procedures.

Exclusion criteria:

* Patients with type 1 diabetes mellitus, gestational diabetes, or diabetes secondary to pancreatic disorders, drug or chemical agent intake.
* Male and female younger than 18 and older than 75 years old.
* Patients with HbA1c ≤7% and ≥9.5%.
* Patients with 20 kg/m^2 > body mass index (BMI) >40 kg/m^2.
* Patients with history of hypersensitivity to metformin.
* Patients with history of hypersensitivity to vildagliptin.
* Lactose intolerance, lactase deficit, glucose-galactose malabsorption.
* Patients who have a history of acute metabolic complications such as lactic acidosis, diabetic pre-coma, diabetic ketoacidosis or hyperosmolar hyperglycemic state within 3 months before study entry.
* Patients who were treated with insulin or glucagon-like peptide-1 (GLP-1) analogue.
* Patients who have been treated by thiazolidinediones (pioglitazone) in the last 6 months.
* Use of systemic glucocorticosteroids (excluding topical application or inhaled forms) for 7 consecutive days or within more than 3 months prior to study entry.
* Patients with impaired hepatic function (alanine transaminase [ALT], aspartate transaminase [AST] activity >1.5 times the upper limit of normal [ULN]).
* Patients with impaired renal function (serum creatinine concentration >135ɥmol/l in men and >110ɥmol/l in female).
* Patients who had experienced myocardial infarction, stroke, unstable angina or coronary artery bypass surgery within 6 months prior to screening, or patients with arrhythmia requiring treatment.
* Patients with chronic heart failure II-IV functional class according to the classification of NYHA (New York Heart Association).
* Patients taking medicines of thyroid hormones, warfarin, dicoumarin or digoxin.
* Patients who took sodium channel blockers and SGLT2 inhibitors (or inhibitors sodium glucose transporters 2) in the last 6 weeks prior to study entry.
* Known history of alcohol or drug abuse within 6 months prior to screening.
* Pregnant or woman during breast feeding period.
* Women of childbearing potential not protected by effective contraceptive method of birth control.
* Men whose partners are planning pregnancy.
* History of hypersensitivity to the study drug or to a drug with a similar chemical structure.
* Use of any investigational drug within 3 months prior to study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Up to Week 24

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | Up to Week 24
Change from baseline in postprandial glucose | Up to Week 24
Percentage of patients achieving HbA1c <7% and <6.5% | Up to Week 24
Percentage of patients with at least one episode of hypoglycemia | Up to Week 24
Number of episode of hypoglycemia (symptomatic, asymptomatic, severe hypoglycemia) | Up to Week 24
Change from baseline in body weight | Up to Week 24
Number of adverse events | Up to Week 24
Number of serious adverse events | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site 03, Vladimir, Vladimirskaya Oblast’, Russia